CLINICAL TRIAL: NCT06383221
Title: A Randomized Controlled Trial of the "Psychological Training Camp & Obstetrician-Led Psychoprenatal Intervention (PICONI)" Stepwise Intervention Model for Depression and Anxiety During Pregnancy.
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Fangbiao Tao (Other)
Responsible Party: Sponsor-Investigator, Fangbiao Tao, Professor, Anhui Medical University
Organization: Anhui Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 83244570
Record Dates: First submitted 2024-04-22; First posted 2024-04-25 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Perinatal Depression; Stepped Care; Perinatal Anxiety

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): Pregnant women with mild anxiety and/or depression self-study the Psychic Fitness Camp, and pregnant women with moderate-to-severe anxiety and/or depression self-study the Psychic Fitness Camp with immediate referral to an obstetrician for one to three Mood Scan.
  Interventions: Combination Product: "Mental Fitness Boot Camp - Advanced Counseling" Step-by-Step Care
- control group (No Intervention): The control group received routine care.

INTERVENTIONS:
Combination Product: "Mental Fitness Boot Camp - Advanced Counseling" Step-by-Step Care — Simple and scientific advice
  Arms: intervention group

SUMMARY:
In this study, pregnant women were screened and managed for depression and anxiety in three time windows: early pregnancy, mid-pregnancy, and late pregnancy. Pregnant women who screened positive for depression and/or anxiety during pregnancy were dynamically enrolled in the study and stratified into randomized groups based on gestation period (early/mid and late), depression and/or anxiety, randomly assigned to the intervention and control groups on a 1:1 basis. Pregnant women with mild anxiety and/or depression self-study the Psychic Fitness Camp, and pregnant women with moderate-to-severe anxiety and/or depression self-study the Psychic Fitness Camp with immediate referral to an obstetrician for one to three Mood Scan. The control group received routine care.

DETAILED DESCRIPTION:
The intervention group used the "Psychological Training Camp & Obstetrician-Led Psychoprenatal Intervention (PICONI)" stepwise care model, which incorporated cognitive-behavioral therapy, mindfulness,etc., with the Psychic Fitness Camp being a self-help learning experience and the Mood Scan being a perinatal clinic doctor guiding pregnant women in unhealthy thinking alternatives and behavior design.

Metabolic markers of perinatal depression anxiety and the mitigating effects of the stepped care model were explored by collecting blood and urine samples from the study participants during early, mid and late pregnancy respectively, samples were collected and stored in a refrigerator at -80 degrees Celsius.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women; Informed consent, able to complete the questionnaire independently; Positive first depression screening (EPDS ≥ 10) or anxiety screening (GAD-7≥5) in early and mid pregnancy; Intention to have children in this pregnancy.

Exclusion Criteria:

* Suffering from depression being treated with psychotherapy or medication

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2024-05-20 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-07-10 (Estimated)

PRIMARY OUTCOMES:
Edinburgh Postnatal Depression Scale | 42 days postpartum
  Assessment of the severity of depressive symptoms

SECONDARY OUTCOMES:
Generalized Anxiety Disorder, Ages and Stages Questionnaires, Maternal Postnatal Attachment Scale | late pregnancy, 42 days postpartum, three months postpartum, six months postpartum
  Assessment of the severity of anxiety symptoms, birth outcome, growth and development in children, Mother-infant attachment relationship
World Health Organization Five-item Well-Being Index | late pregnancy, 42 days postpartum
  Assessment of the Well-Being index

CONTACTS AND LOCATIONS:
Locations (1):
- Ma'anshan Maternal and Child Health Center, Ma’anshan, China

IPD SHARING:
Plan to Share IPD: Undecided